CLINICAL TRIAL: NCT07404332
Title: Phase I Study of 5-Azacitidine Plus PD-1/PD-L1 Inhibitor in Patients With PD-1/PD-L1 Refractory Tumors
Brief Title: 5-Azacitidine Plus PD-1/PD-L1 Inhibitor With PD-1/PD-L1 Refractory Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mohammed Milhem (Other)
Responsible Party: Sponsor-Investigator, Mohammed Milhem, Clinical Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202511023
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumor; Locally Advanced Solid Tumor; Metastatic Tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Azacitidine; pembrolizumab; Nivolumab; cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 5-Azacitidine Plus PD-1/PD-L1 inhibitor (Experimental): This Phase I study will assess 6 doses of 5-Azacitidine (5, 10, 15, 25, 50 and 75 mg/m2) in combination with a PD1/PD-L1 inhibitor. The PD1/PD-L1 inhibitor will be given at standard of care dosing approved by the FDA for this indication. Inhibitors approved for study indications include Pembrolizumab, Nivolumab, and Cemiplimab.
  Interventions: Drug: 5 Azacytidine; Drug: Pembrolizumab; Drug: Nivolumab; Drug: Cemiplimab

INTERVENTIONS:
Drug: 5 Azacytidine — 5-Azacitidine (Azacitidine) is a nucleoside analogue chemotherapy drug
Drug: Pembrolizumab — Pembrolizumab is a high-affinity humanized monoclonal antibody that functions as immune checkpoint inhibitor
Drug: Nivolumab — Nivolumab is a high-affinity humanized monoclonal antibody that functions as immune checkpoint inhibitor
Drug: Cemiplimab — Cemiplimab is a high-affinity humanized monoclonal antibody that functions as immune checkpoint inhibitor

SUMMARY:
This is a Phase I study to determine the optimal biological dose (OBD) of 5-Azacitidine in combination with PD-1/PD-L1 inhibitors in patients with tumors refractory to PD-1/PD-L1 inhibitors, for which such treatments have been approved.

DETAILED DESCRIPTION:
This is a Phase I study to determine the optimal biological dose (OBD) of 5-Azacitidine in combination with PD-1/PD-L1 inhibitors in patients with tumors refractory to PD-1/PD-L1 inhibitors, for which such treatments have been approved.

This Phase I study will assess 6 doses of 5-Azacitidine (5, 10, 15, 25, 50 and 75 mg/m2) in combination with a PD1/PD-L1 inhibitor. The PD1/PD-L1 inhibitor will be given at standard of care dosing approved by the FDA for this indication.

ELIGIBILITY:
Inclusion Criteria:

* Written and voluntary informed consent.
* At least 18 years of age or older.
* Histologically and radiologically confirmed locally advanced or metastatic unresectable solid tumor malignancy for which PD-1 or PD-L1 therapy is already approved by the FDA. Locally advanced is defined as unresectable in the opinion of the treating physician. A repeat biopsy is required if previous biopsy tissue is unavailable.
* At least one Response Evaluation Criteria in Solid Tumors (RECIST 1.1) - defined target lesion.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 (fully active, able to carry on all pre-disease performance without restriction), 1 (restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, such as light housework or office work), or 2 (ambulatory and capable of self-care but unable to carry out any work activities, spending more than 50% of waking hours up and about).
* Documented progression on PD1 or PD-L1 inhibitors.
* Recovery from any acute toxicity associated with prior therapy to grade 1.
* Renal function (creatinine level within normal institutional limit, or creatinine clearance >15 mL/min/1.73 m2 for patients with creatinine levels above institutional normal, calculated using the Cockcroft-Gault formula).
* Liver function (AST/ALT <3.0 X institutional upper limit of normal OR <5 X institutional upper limit of normal in cases of liver metastasis; total bilirubin ≤ 1.5 times upper limit of normal).
* Adequate hematological lab values including:

  * Absolute Neutrophil Count (ANC) ≥ 1.0 X 109/L
  * Platelets ≥ 100X109/L
  * Hemoglobin ≥ 7.0 g/dL
* Female subjects of childbearing potential and non-sterilized male subjects who intend to be sexually active during the study must agree to use a highly effective method of contraception from time of screening, throughout the whole duration of the drug treatment, and during the 6-month post-treatment washout period.
* Patients may have previously received a hypomethylating agent, as long as it was not given in combination with ipilimumab.
* Patients may have previously received ipilimumab but must have relapsed or progressed while on therapy.
* Patients must have adequate archival tissue available for the purpose of downstream methylation status assessment, immunohistochemistry, RNA expression (10 slides at 5µM). If archival tissue is not available, a repeat biopsy is required.

Exclusion Criteria:

* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen.
* Patients with active, untreated metastases in the central nervous system.
* Patients who are pregnant or breastfeeding.
* Patients who have an active infection.
* Patients with significant hematologic, hepatic, and renal function impairment.
* Patients who are being treated for any concurrent medical condition requiring the use of systemic steroids or history of long-term use of systemic steroids.
* Patients who have a history of inflammatory bowel disease or a history of symptomatic autoimmune disease.
* Patients who have had any major surgical procedure or significant traumatic injury within 28 days prior to study enrollment.
* Patients who have received chemotherapy, immunosuppressive agents or any investigational drug within 28 days prior to starting the study drugs.
* Patients who have any underlying medical condition which, in the treating physician's opinion, will make the administration of study drugs hazardous or obscure the interpretation of adverse events.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities and responses as defined by CTCAE v5.0 | Treatment initiation through 30 days +/- 7 days post completion of therapy
  Assess the safety and tolerability of 5-Azacitidine Plus PD-1/PD-L1 inhibitor

SECONDARY OUTCOMES:
Proportion of participants with a complete response (CR) | Treatment initiation through five years
  The proportion of patients with a pathologic complete response, defined as disappearance of all target lesions, disappearance of all non-target lesions and normalization of tumor marker level
Proportion of participants with a partial response (PR) | Treatment initiation through five years
  At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD
Overall Survival (OS) | Treatment initiation through five years
  Time from study treatment initiation to death due to any cause
Progression Free Survival (PFS) | Treatment initiation through five years
  Time from study treatment initiation to disease progression or death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Milhem, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Health Care, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No